CLINICAL TRIAL: NCT02323347
Title: Cut-Off Progesterone Values Deleterious for In Vitro Fertilization and Fresh Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Dr. Francisca Martínez, PhD, Fundacion Dexeus
Other Study IDs: PROGEDEX2014
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Progesterone; Fertilization in Vitro; Infertility; Pregnancy
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Progesterone — Progesterone level

SUMMARY:
At which deleterious cut off value of progesterone on day of HCG (P-hCG) in our IVF program should fresh embryo transfer (ET) be cancelled?

DETAILED DESCRIPTION:
There is still an ongoing debate on the effect of subtle increased P-hCG concentration on pregnancy outcome after fresh ET. No consensus on the cut-off value to define increased P-hCG seems to exist. It is accepted that high P advances endometrium, leading to asynchrony between the implanting embryo and the endometrium, and resulting in implantation failure. A freeze all embryos policy and postponement of ET in subsequent frozen-thawed cycle has been proposed.

ELIGIBILITY:
Inclusion Criteria:

* Fresh embryo transfer
* Progesterone value on day HCG (Human choriogonadotrophin hormone)

Exclusion Criteria:

* Clinical indication for delaying embryo transfer

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing IVF-ICSI ad fresh embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 1901 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy | 6 weeks after embryo transfer procedure

REFERENCES:
- [Derived] Martinez F, Rodriguez I, Devesa M, Buxaderas R, Gomez MJ, Coroleu B. Should progesterone on the human chorionic gonadotropin day still be measured? Fertil Steril. 2016 Jan;105(1):86-92. doi: 10.1016/j.fertnstert.2015.09.008. Epub 2015 Oct 9. PMID 26453983